CLINICAL TRIAL: NCT05231499
Title: Host Immunity and Nasal Fungal Colonization
Brief Title: Immunity and Nasal Fungal Colonization
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE18237B
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Colonization, Asymptomatic
Keywords: colonization; microbiota; fungi; immunocompromised
MeSH Terms: conditions — Asymptomatic Infections | interventions — Nasal Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers
- immunocompromised subjects
  Interventions: Other: nasal irrigation

INTERVENTIONS:
Other: nasal irrigation — regular saline nasal rinse
  Groups: immunocompromised subjects

SUMMARY:
Fungal colonization causes opportunistic infection that may manifest when the host's immune status deteriorates. The purpose of this study was to determine the prevalence of fungal colonization in immunocompromised subjects compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised subjects included those who had known risk factors for fungal infection, including malignant diseases, diabetes, autoimmune disorders, renal or hepatic insufficiency, organ transplantation, or use of immunosuppressants
* Healthy volunteers had neither sinonasal symptoms nor nasal endoscopic inflammation.

Exclusion Criteria:

* Patients were excluded if they were under 20 years old, were receiving antifungal medication, or were pregnant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Immunocompromised subjects have rhinosinusitis or not using nasal irrigation or not using nasal irrigation
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
nasal lavage pooled fungal microbiota | 1 month

SECONDARY OUTCOMES:
nasal lavage aspergillus qPCR | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology, Taichung Veterans General Hospital, Taichang, Taiwan

IPD SHARING:
Plan to Share IPD: No